CLINICAL TRIAL: NCT01570114
Title: EFFICACY OF A SELF EXPANDABLE FULLY COVERED METALLIC STENT IN THE TREATMENT OF BENIGN COLONIC STRICTURES
Brief Title: Covered Metallic Stent and Benign Colonic Strictures
Status: Completed | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, VANBIERVLIET, Medical doctor - study coordinator and director of the endoscopy unit in universitary hospital of Nice (France), Société Française d'Endoscopie Digestive
Other Study IDs: FCSEMS
Record Dates: First submitted 2012-03-29; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-03

CONDITIONS: Colonic Diseases; Stricture; Occlusion
Keywords: Covered metallic stent; colon; benign stricture
MeSH Terms: conditions — Colonic Diseases; Constriction, Pathologic; Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- covered metallic stent: Endoscopically insertion of fully covered metallic stent on benign colonic strictures
  Interventions: Device: Fully covered metallic colonic stent

INTERVENTIONS:
Device: Fully covered metallic colonic stent — Endoscopically insertion of fully covered metallic colonic stent

SUMMARY:
Self-expanding metallic stent placement is a safe and effective endoscopic procedure increasingly used to relieve colonic obstruction. Fully covered metal stents (FCSEMS) and plastic stents have been recently developed to reduce both hyperplastic (non tumoral) and tumoral tissue ingrowth. These fully covered metal or plastic stents have several advantages over non-covered stents, including the possibility of retrieval and limited local tissue reaction, while providing alleviation of obstruction at possibly lower costs. Only few reports of fully covered metal stent placement in patients with benign colorectal strictures are available in the literature. The aim of this study was to assess the effectiveness of FCSEMS in the management of the colonic benign strictures.

DETAILED DESCRIPTION:
It is a national multicentric retrospective study on the use of fully covered metal stent placement in patients with benign colorectal strictures.

Consecutive patients above 18 years of age with a symptomatic benign colonic stricture despite optimal medical and/or endoscopic dilation therapy and which required the use of a FCSEMS were included. All strictures were confirmed to be benign by histology. All details concerning previous history, origins and treatment (medical or endoscopic) of the colonic stenosis were collected from the medical file.

Senior endoscopists with an experience of more than 50 colonic stent placements performed the procedure under general propofol-induced anesthesia with the same technic (The stent was placed under fluoroscopic and videoendoscopic controls).

Patients were required after the procedure to take oral osmotic laxatives regularly. Post-stenting complications were defined as immediate (during the procedure), early (occurring ≤ 30 days) and late (> 30 days) after the procedure. Stent removal and routine follow up endoscopy were scheduled 4 to 6 weeks after placement in most patients or earlier if complications occurred.

All patients were followed up at regular intervals based on their clinical situation. A retrospective chart review was performed to analyze the long-term outcome of the patients.

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 years of age
* symptomatic benign colonic stricture despite optimal medical and/or endoscopic dilation therapy

Exclusion Criteria:

* Previous insertion or treatment of the stricture with metallic (covered or uncovered) stent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in universitary tertiary care center benefited from a fully covered metallic colonic stent for treatment of benign stricture
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Symptom resolution of colonic occlusion | 48 hours
  Defined as the clinical (stools, stop pain) and radiological evidence of colonic decompression within 48 hours of stent insertion and without the need for reintervention

SECONDARY OUTCOMES:
Successful stent placement | Immediatly after stent insertion (one minute)
  On the first attempt with complete deployment and precise positioning of the stent at the location of the stenosis, which was confirmed by fluoroscopy
Successful stent retrieval | One minute (during colonoscopy for stent retrieval)
  Possibility of retrieval the stent with a snare or a forceps
Occurrence of any complication during interventional endoscopy, stent retrieval and the follow-up | 60 days
  Perforation, bleeding, migration, pain, fecal incontinence and foreign body sensation, stent impaction and hyperplastic tissue overgrowth
Recurrence of colonic occlusion | 60 days, 6 months and one year
  New episode of occlusion or subocclusion (pain with stool and gas discontinuation and imaging with cecum dilation) after stent retrieval or migration

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy Vanbiervliet, MD, Principal Investigator — Société Française d'Endoscopie Digestive